CLINICAL TRIAL: NCT03906409
Title: Effect of Nutrient Delivery Pattern on Biological Rhythms in Human Skeletal Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, James Betts, Professor James Betts, University of Bath
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FE
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Circadian Rhythms; Feeding Patterns
Keywords: Feeding Patterns; Skeletal Muscle; Metabolism; Circadian Rhythms; Diurnal Rhythms
MeSH Terms: conditions — Feeding Behavior | interventions — NOP-bolus regimen

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to one of two parallel trial arms: constant feed or bolus feed
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constant (Active Comparator): Participants will be provided with their daily energy requirements in a continuous drip across the day (1 ml/minute).
  Interventions: Other: Constant
- Bolus (Experimental): Participants will be provided with their daily energy requirements in two bolus feeds. One at 08:00-08:15 and one at 20:00-20:15
  Interventions: Other: Bolus

INTERVENTIONS:
Other: Constant — Participants will be provided with their daily energy requirements in a continuous drip across the day (1 ml/minute).
  Arms: Constant
Other: Bolus — Participants will be provided with their daily energy requirements in two bolus feeds. One at 08:00-08:15 and one at 20:00-20:15
  Arms: Bolus

SUMMARY:
Recent work has established biological rhythms in human skeletal muscle. It remains unknown how the timing and pattern of meals influences these rhythms. Therefore, this study sets out to establish how frequent (CONSTANT) vs infrequent (BOLUS) feeding patterns influence established biological rhythms in skeletal muscle.

DETAILED DESCRIPTION:
Human metabolism is regulated on a daily basis via a circadian timing system that coordinates metabolic responses between various tissues. Skeletal muscle is a major site for the oxidation or storage of key metabolites, with recent studies at Bath and Surrey demonstrating biological rhythms in this tissue over a 24-h cycle. It is well established that dysregulated metabolism in skeletal muscle contributes to poor metabolic health and that poor diet is a causal factor in this deterioration. Diet can be characterised by three nutritional considerations: how much is eaten (i.e. quantity/dose), what is eaten (i.e. type) and when it is eaten (i.e. timing). Whilst most dietary approaches and most scientific studies have focused on the first two factors, there is convincing evidence that human health is also dictated by the pattern of nutrient delivery; this includes the frequency and regularity of daily eating occasions, along with their timing both in absolute terms (i.e. time-of-day) and relative to when other inter-related daily events occur - or usually occur (e.g. light exposure, sleep, exercise, etc.).

It remains unknown whether the interaction of such factors may affect the biological rhythms previously documented in human skeletal muscle. In particular, from a basic science perspective, the fundamental contrast between frequent versus infrequent feeding warrants investigation. To this end, 16-24 healthy adults will be randomly allocated to receive their individual daily energy requirements delivered via naso-gastric infusion either continuously over 24 hours (n=8-12; CONSTANT) or as two bolus infusions at the start (0800 h) and mid-point (2000 h) of the monitoring period (n=8-12; BOLUS). Serial skeletal muscle (vastus lateralis) biopsies will be sampled every 4 hours over a controlled 24-h sleep-wake cycle.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index >19 but <30 kg/m2
* Be able and willing to give informed oral and written consent, complete and meet the defined criteria of pre-study questionnaires and screens,
* Have a regular sleep cycle with a sleep duration between 6 and 8 hours, do not exhibit extreme morning or evening preference (Horne and Ostberg, 1976)
* Agree to keep a constant sleep/wake cycle with a self-selected 8 hour sleep duration (from which it cannot be deviated by more than 30 minutes) for one week prior to the lab study,
* Obtain 15 minutes of sunlight within 1.5 hours of waking up and agree to nap only within a 4 h designated nap window for one week prior to the lab study,
* Allow confirmation of compliance to these instructions by wearing ActiHeart monitors continuously and complete daily sleep and event diaries for one week before the study session,
* Agree to refrain from alcohol, caffeine, heavy exercise and certain food components TWO days before the study session,
* Agree to weigh and record daily meals (based on individual energy requirements) for TWO days prior to the study,
* Agree to refrain from prescribed and 'over the counter' medication and food/vitamin supplements for a wash-out period three weeks before and during the study.

Exclusion Criteria:

* Are taking regular medication (also non-prescribed) or food supplements (e.g vitamins, minerals, fish oil, antioxidant tablets) from which it is not possible to refrain, known to influence: Sleep/alertness/the circadian timing system (e.g beta-blockers, barbituates, antidepressants, benzodiazepines, melatonin, ritalin, modafinil, soporifics, St John's Wort), any of the metabolic functions (e.g. affecting thyroid, kidney, liver or gastrointestinal function)
* Any of the inflammatory markers (e.g. aspirin, ibuprofen, antiobiotics, hay fever medication, medication for sore throats and colds)
* And/or any of the endothelial markers (e.g. ACE inhibitors and angiotensin (receptor) blockers, diuretics, Beta-blockers, anti-thrombosis medication),
* Have a history of any circadian or sleep disorder or metabolic, cardiovascular or chronic infectious / inflammatory disease as confirmed by the GP or the pre-study questionnaires (e.g. a Pittsburgh Sleep Quality Index > 5 will result in exclusion),
* Have a history of psychiatric or neurological disease or drug and alcohol abuse,
* Have donated over 400 ml of blood in the three months preceding the study,
* Have participated in shift work or have travelled across more than two time zones within three weeks of the study,
* Do not keep a regular sleep-wake cycle,
* Do not refrain from alcohol, caffeine containing drinks (e.g. coffee, coke, tea, redbull), heavy exercise and certain foods (e.g. those high in fat and green vegetables) TWO days before and during the laboratory session,
* Normally consume more than 4 cups of caffeinated beverages (e.g. tea, coffee, cola) daily
* Smokers

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Autophagy | 4 hours
  Rhythms in autophagy with different feeding patterns
Transcriptomic, rhythms in human skeletal muscle | Over a 24-hour period at a 4 hour resolution
  Assessing rhythms in core-clock genes within the muscle samples

SECONDARY OUTCOMES:
Endocrine responses of systemic blood plasma over 24-hours | 24-hours
  Rhythms in endocrine regulation of metabolism over a 24-hour period (e.g. insulin, appetite hormones)
Continuously monitored subcutaneous interstitial glucose concentrations | 48-hours
  Assessed using a continual glucose monitor

CONTACTS AND LOCATIONS:
Overall Officials: Harry A Smith, MSci, Principal Investigator — University of Bath; James A Betts, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Christou S, Wehrens SMT, Isherwood C, Moller-Levet CS, Wu H, Revell VL, Bucca G, Skene DJ, Laing EE, Archer SN, Johnston JD. Circadian regulation in human white adipose tissue revealed by transcriptome and metabolic network analysis. Sci Rep. 2019 Feb 25;9(1):2641. doi: 10.1038/s41598-019-39668-3. PMID 30804433
- [Background] Perrin L, Loizides-Mangold U, Chanon S, Gobet C, Hulo N, Isenegger L, Weger BD, Migliavacca E, Charpagne A, Betts JA, Walhin JP, Templeman I, Stokes K, Thompson D, Tsintzas K, Robert M, Howald C, Riezman H, Feige JN, Karagounis LG, Johnston JD, Dermitzakis ET, Gachon F, Lefai E, Dibner C. Transcriptomic analyses reveal rhythmic and CLOCK-driven pathways in human skeletal muscle. Elife. 2018 Apr 16;7:e34114. doi: 10.7554/eLife.34114. PMID 29658882